CLINICAL TRIAL: NCT06743633
Title: An Observational Study to Explore the Association Between Beta Blocker Use and Depressive Outcomes
Brief Title: Association of Beta Blocker Use with Depressive Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Chitkara University (Other)
Responsible Party: Sponsor
Other Study IDs: 2350981060
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Depression - Major Depressive Disorder
Keywords: Beta-blockers; Depression; Prevalence
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Prospective study: Cardiovascular disease patients on β-blockers therapy atleast from last 1 year: Evaluation of depression status using ICD 10, HADS, PHQ-9
- Prospective study: Cardiovascular disease patients without β-blockers therapy: Evaluation of depression status using ICD 10, HADS, PHQ-9.
- Retrospective study: Clinically diagnosed Depression patients + Cardiovascular comorbidities: To determine the prevalence of patients on β-blocker use among clinically diagnosed depression patients with cardiovascular comorbidities by reviewing their medical records.
- Retrospective study:Clinically diagnosed Depression + Cardiovascular comorbidities without β-blocker: To determine the prevalence of patients without β-blocker use among clinically diagnosed depression patients with cardiovascular comorbidities by reviewing their medical records.

SUMMARY:
An Observational Study to Explore the Association Between β-Blocker Use and Depressive Outcomes

DETAILED DESCRIPTION:
Study design- This is a Prospective, Retrospective, Cross-sectional observational study. In prospective study, cardiovascular patients will be divided into two groups: those taking β-blockers and those not taking β-blockers. A questionnaire-based study will be conducted to assess the depression status of both groups. The study will include Depression Inventory (MDI) (lCD-10), Hamilton Rating Scale for Depression (HDRS) and Patient health questionnaire-9 (PHQ-9) for prospective study.

In the Retrospective study, clinically diagnosed depression patients with cardiovascular co morbidity will be identified from the psychiatric department.

Study population- Total number of patients to be included in both prospective and retrospective study: 1136 Prospective: 684 participants from cardiology department (two subgroups = 342 with β-blockers and other 342 without β-blockers) Retrospective: 452 participants from psychiatric department (two subgroups = 226 with β-blockers and other 226 without β-blockers) Planned time period for the study: Jan 2025 to May 2025 Procedure- Prospective: A prospective study, a total of 684 cardiovascular participants will be recruited from the Cardiology department. Participants will be divided into two groups: participants who are currently on β-blockers from at least 1 year and those who are not on β-blockers. Then a Depression Inventory (MDI) (lCD-10), Hamilton Rating Scale for Depression (HDRS) and PHQ-9 (Patient health questionnaire-9) depression questionnaire will be run on both to assess depression levels. Data collected from both groups will be compared to evaluate differences in depression status.

Retrospective: A retrospective study will be conducted involving 452 patients diagnosed with depression and atleast one cardiovascular co morbidity from the psychiatry department. Patients will be classified into two groups: those who were prescribed with β-blockers and those who were not. Medical records of these patients will be obtained from their respective Staff. The primary objective is to determine the prevalence of β-blocker use among depressed patients with cardiovascular conditions by reviewing their medical histories.

ELIGIBILITY:
For Prospective Study:-

Inclusion Criteria:

1. Participants aged from ≥18 years at the time of consent.
2. Participants on β-blockers for at least 1 year.
3. No significant cognitive impairment.
4. Participants who are willing to participate.
5. To be able to understand and answer the self-assessment questionnaires.

Exclusion Criteria:

1. Having severe sensory and physical limitations, severe disconnection from the environment, or presence of severe neuropsychiatric symptoms that make it impossible to administer the assessment.

For Retrospective Study:-

Inclusion criteria:

1. Diagnosis with major depressive disorder or reference to "clinical depression" in patient charts.
2. Participants with cardiovascular co-morbidity.
3. Participants aged from ≥18 years.

Exclusion criteria:

1. Depression with other psychiatric illness for e.g., schizophrenia, cognitive impairment and without any cardiac comorbidity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total number of patients to be included in both prospective and retrospective study: 1136 Prospective: 684 participants from cardiology department (two subgroups = 342 with β-blockers and other 342 without β-blockers) Retrospective: 453 participants from psychiatric department (two subgroups = 226 with β-blockers and other 226 without β-blockers)
Sampling Method: Probability Sample
Enrollment: 1136 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
An Observational Study to Explore the Association Between β-Blocker Use and Depressive Outcomes | 6 months
  β-blockers use are associated with antidepressant effect or not

IPD SHARING:
Plan to Share IPD: No